CLINICAL TRIAL: NCT06628674
Title: Developing and Testing the Effect of Online Interactive Videos in Improving Low Anterior Resection Syndrome, Psychological Distress,and Quality of Life
Brief Title: Developing and Testing the Effect of Online Interactive Videos in Improving Low Anterior Resection Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202301931B0
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-08

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Core muscle exercise (Experimental)
  Interventions: Behavioral: core muscle exercise
- pelvic muscle exercise (Other)
  Interventions: Behavioral: pelvic muscle exercise

INTERVENTIONS:
Behavioral: core muscle exercise — Patients in experiment group will do core muscle exercise with online interactive videos
  Arms: Core muscle exercise
Behavioral: pelvic muscle exercise — Patients in experiment group will do pelvic muscle exercise without online interactive videos
  Arms: pelvic muscle exercise

SUMMARY:
This study aims to develop and test the effect of online interactive videos in improving LARS.

ELIGIBILITY:
Inclusion Criteria:

1. Stage I-III rectal cancer.
2. Patients already know their condition.
3. Aged 20 years and older.
4. Consciously communicate in Mandarin or Taiwanese.
5. Agreed with the interview and had signed the permit.

Exclusion Criteria:

1. Recurrent rectal cancer.
2. Stage IV rectal cancer.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Self-report Questionnaire | Change from baseline symptom to 6 months after intervention
  Show the specific trajectory of LAR Syndrome, psychological distress and fecal incontinence-related QoL in patients with rectal cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan District, 中和區, Taiwan